CLINICAL TRIAL: NCT03275558
Title: Phase I Clinical Trial of Nasal Spray in Treating Patients With Recurrent Glioblastoma, Gliosarcoma, Glioma
Brief Title: Clinical Trial of the Use of the Nasal Spray of Patients With Recurrence of Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prior to enrollment of first participant. (It has been determined on 2018 May 15 that the NCT03275558 study will be stopped by sponsor decision)
Sponsor: Center Trials & Treatment (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NST-4-G
Record Dates: First submitted 2017-08-30; First posted 2017-09-07 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Glioblastoma; Gliosarcoma; Anaplastic Gliomas
Keywords: Nasal Spray; Gliosarcoma; Glioblastoma; Gliomas
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — Axitinib; Sunitinib; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Axitinib (Active Comparator): A single dose of Axitinib - 1 mg in a liquid form in the composition (Axitinib+Sunitinib+Pazopanib) of the nasal spray.
  Interventions: Drug: Axitinib 1 MG
- Sunitinib (Active Comparator): A single dose of Sunitinib- 5 mg in a liquid form in the composition (Axitinib+Sunitinib+Pazopanib) of the nasal spray.
  Interventions: Drug: Sunitinib 5 MG
- Pazopanib (Active Comparator): A single dose of Pazopanib-5 mg in a liquid form in the composition (Axitinib+Sunitinib+Pazopanib) of the nasal spray.
  Interventions: Drug: Pazopanib 5 MG

INTERVENTIONS:
Drug: Axitinib 1 MG — Pharmaceutical composition of Axitinib 5MG +Sunitinib 5MG + Pazopanib 5MG in the liquid form of a nasal spray NST-4-G.
  Subjects take a nasal spray BID at a single dose in each nostril (approximately at the same time of day) for 7 weeks or unacceptable toxicity or other adverse events.
  Other Names: AG 013736, Inlyta
  Arms: Axitinib
Drug: Sunitinib 5 MG — Pharmaceutical composition of Axitinib 5MG +Sunitinib 5MG + Pazopanib 5MG in the liquid form of a nasal spray NST-4-G.
  Other Names: SU11248, Sutent
  Arms: Sunitinib
Drug: Pazopanib 5 MG — Pharmaceutical composition of Axitinib 5MG +Sunitinib 5MG + Pazopanib 5MG in the liquid form of a nasal spray NST-4-G.
  Other Names: GW786034, Votrient
  Arms: Pazopanib

SUMMARY:
This is a study to determine the efficacy, safety and clinical benefit (how well the drugs works), of the pharmaceutical compositions in Nasal Spray NST-4G for the treatment of brain tumors( Recurrent Glioblastoma, Gliosarcoma,Anaplastic Gliomas, Previously Treated).

All drugs target the inhibition of the growth factors and neo-angiogenesis as one the main reasons for the growth of the tumor.

The purpose of the Nasal Spray NST-4G study is to determine the safety and tolerability in order to establish the best dose level to be used in future studies.

DETAILED DESCRIPTION:
This is an open-label study, Phase 1 study evaluating the preliminary safety, efficacy, tolerability and clinical benefit of Nasal Spray NST-4G in patients with Recurrent Glioblastoma, Gliosarcoma,Anaplastic Gliomas.

Acceptable subjects included in the study will receive Nasal Spray NST-4G, administered twice daily for 7 weeks intranasally.

Every 8th day, a blood function (hematopoiesis) is examined . Patients may continue to receive subsequent nasal spray cycles if the subject is not intolerant of the test product, does not withdraw consent or the individual no longer receives clinical benefit (the factors taken for consideration will be the progression of the disease, expressed in increasing neuropathy, hemiparesis, pain intensification ,DLT events, Clinical signs of deteriorating quality of life (QOL).

The evaluation of the tumor size will be repeated using the MRI method with a contrast agent after each 7-week nasal spray cycle.

The use of nasal spray is a non-invasive method of treatment that does not require specialized conditions for therapy

ELIGIBILITY:
Inclusion Criteria:

1. Has been treated previously with bevacizumab and (or) temozolomide.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be >/= 18 years of age on day of signing informed consent.
4. Have histologically confirmed World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma). Participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made.
5. Patients must be at first or second relapse and clinically require reoperation for tumor progression within 4 to 6 weeks. Note: Relapse is defined as progression following initial therapy (i.e., radiation, chemotherapy, or radiation+ chemotherapy). If the participant had a surgical resection for relapsed disease and no antitumor therapy instituted for up to 12 weeks, this is considered one relapse. For participants who had prior therapy for a low grade glioma, the surgical diagnosis of a high grade glioma will be considered first relapse.
6. Have measurable disease consisting of a minimal volume of 1 cm3.
7. Have provided tissue from an archival tissue sample of a tumor lesion.
8. Have a performance status of >/= 60 on the KPS.
9. Stable dose of steroids for 5 days, no more than 2 mg dexamethasone (or equivalent) total per day
10. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days prior to registration. 1) Hematological : Absolute neutrophil count (ANC) >/=1,500 /mcL; Platelets >/=100,000 / mcL; Hemoglobin >/= 9 g/dL or >/= 5.6 mmol/L. 2) Renal: Serum creatinine </= 1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) >/= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN.
11. Hepatic: Serum total bilirubin </= 1.5 X ULN OR Direct bilirubin </= ULN for subjects with total bilirubin levels > 1.5 ULN; AST (SGOT) and ALT (SGPT) </= 2.5 X ULN, Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) </= 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) </= 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
12. Female subject of childbearing potential should have a negative serum pregnancy test.
13. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 90 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy.

Exclusion Criteria:

1. Has tumor localized primarily to the brainstem or spinal cord.
2. There are acute or chronic diseases of the maxillary and paranasal sinuses, sphenoid sinuses, the sinuses of the trellis, early or current traumatic injuries of these zones, fractures of the nasal septum, congenital malformations of the development of bone tissue of the latticed bone.
3. Is currently participating in or has participated in a study of an investigational agent or using an investigational device 4 weeks since last dose of agent administration.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 2 mg of dexamethasone total per day or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
5. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Subjects with alopecia, </= Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has known carcinomatous meningitis, extracranial disease, or multifocal disease.
9. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study.
10. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known history of Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
The definition of survival without progression of disease | From the date of commencement of participation in the study until the date of first documented progression or date of death from any cause, whichever came first /assessed up to 48 months/
  The definition of survival without progression of disease is estimated as time of the disease-free period / absence of continued tumor growth (in weeks) by objective methods of control (MRI or CT)

SECONDARY OUTCOMES:
The definition of overall survival | From the date of commencement of participation in the study until date of death from any cause / assessed up to 60 months/
  The determine overall survival from the date of commencement of participation in the study until date of death from any cause.
The definition late toxicity to maximum tolerated dose (MTD) | From the date of commencement of participation in the study until the onset of adverse event /assessed up to 48 months/
  To determine late toxicity for the maximum tolerated dose is estimated a function of hematopoiesis of patients by blood sampling every 8th day The MTD is based upon dose-limiting toxicities (DLTs) experienced during Cycle 1 of treatment. The MTD is the dose level at which 0/6 or 1/6 patients experience DLT with at least two patients experiencing DLT at the next higher dose level. Using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, DLTs are defined as: Grade 4 neutropenia lasting greater than 5 days; Grade 3 thrombocytopenia; the occurrence of non-hematologic Grade 3 or greater drug-related adverse events excluding Grade ≥ 3 elevation in alkaline phosphatase, Grade ≥ 3 nausea or vomiting unless occurring despite the use of standard anti-emetics or Grade 3 diarrhea unless occurring despite standard anti-diarrheal therapy; > 14 day delay to re-treat due to failure to resolve drug-related toxicity to re-treatment criteria or pre-treatment baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Reznic, PhD, Principal Investigator — Center Trials & Treatment Inc.; Oliever R Kolb, Study Director — Center Trials & Treatment Inc.
Locations (2):
- The Hong Kong Cancer Institute, Hong Kong, Hong Kong
- National University Cancer Institute,, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IB, SAP. ICF E-mail: info@trials.clinic
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after September 30, 2017
Access Criteria: On request
URL: https://trials.clinic/